CLINICAL TRIAL: NCT04244604
Title: The Effects of a High Salt Meal on Blood Flow Regulation
Brief Title: Vascular Effects of Acute Sodium (VEAS) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: University of Delaware (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Austin Robinson, Associate Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 23319; K01HL147998 (NIH)
Record Dates: First submitted 2019-12-05; First posted 2020-01-28 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Sodium Excess; Racial Disparities; Blood Pressure; Cardiovascular Risk Factor
Keywords: blood pressure; racial disparities; cardiovascular health; physical fitness; sleep; dietary sodium; dietary salt; diet
MeSH Terms: conditions — Hypernatremia | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The intervention is to provide subjects with either a low sodium meal (140 mg sodium) and a high sodium meal (2500 mg sodium), in a randomized order.
Who Masked: Investigator
Masking Description: The experimenter will be blinded to what sodium condition the participant is in, and all data analysis will be conducted blinded to the condition as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Sodium Meal (2500 mg sodium), Then Low Sodium Meal (140 mg sodium) (Experimental): On experimental visit days, participants will consume each of the experimental meals, in this order. Prior to, and at several timepoints after consumption, they will have sympathetic nerve activity, vascular function, blood pressure and blood samples (from intravenous catheters) assessed.
  Interventions: Other: Low Sodium Meal (140 mg sodium chloride); Other: High Sodium Meal (2500 mg sodium chloride)
- Low Sodium Meal (140 mg sodium), then High Sodium Meal (2500 mg sodium) (Experimental): On experimental visit days, participants will consume each of the experimental meals, in this order. Prior to, and at several timepoints after consumption, they will have sympathetic nerve activity, vascular function, blood pressure and blood samples (from intravenous catheters) assessed.
  Interventions: Other: Low Sodium Meal (140 mg sodium chloride); Other: High Sodium Meal (2500 mg sodium chloride)

INTERVENTIONS:
Other: Low Sodium Meal (140 mg sodium chloride) — Varied amounts of salt (sodium chloride) will be added to a very low sodium soup to determine the effects of a single high sodium meal on measures of vascular function and autonomic regulation of blood pressure. The Low Sodium soup will serve as the control condition.
Other: High Sodium Meal (2500 mg sodium chloride) — Varied amounts of salt (sodium chloride) will be added to a very low sodium soup to determine the effects of a single high sodium meal on measures of vascular function and autonomic regulation of blood pressure. The Low Sodium soup will serve as the control condition.

SUMMARY:
This IRB will cover a current clinical trial (NCT04244604) that was started at Auburn University (AU IRB#19-390), the Principal Investigator's prior institution, and is supported by his NIH Career Development Award (NHLBI K01HL147998).

About nine out of ten Americans overconsume dietary salt. Compared to other racial groups, Black individuals are more prone to salt-sensitive hypertension and negative cardiovascular conditions associated with high salt intake. However, there is a critical need to determine the reasons behind and mechanisms that contribute to these racial disparities. Both acute (single meal) and chronic high-dietary sodium cause small but important increases in blood sodium concentration that are associated with altered blood pressure regulation and blood vessel dysfunction. However, racial differences in these measures have not been examined. This is important because Black individuals generally exhibit lower circulating concentrations of hormones (e.g., renin, aldosterone, angiotensin 2) that buffer changes in body sodium to regulate blood pressure, and this could make them more vulnerable to the negative effects of a high-sodium meal.

Therefore, the purpose of this study is to determine whether there are racial differences in blood pressure regulation and blood flow after a high-sodium meal. The investigators will assess blood pressure regulation, blood vessel stiffness, and the blood vessel's ability to dilate before and after a high-salt meal and a low-salt control meal (both meals are low-salt tomato soup with varied added salt). The investigators will also collect blood and urine to measure sodium and determine biochemical changes that may be contributing to racial differences in cardiovascular function.

DETAILED DESCRIPTION:
The investigators have previously used a high-sodium saline infusion to increase blood sodium and consequently increase blood pressure in Black and White individuals. The investigators' prior data suggest that increased blood sodium concentrations result in larger blood pressure elevations for a given elevation in blood sodium levels in Black compared to White adults. In this proposal, the investigators are seeking to translate these previous findings using a single high-salt meal (up to 2500 mg of sodium; similar to a few slices of pizza or a sandwich/burger and side dish). Our primary aims are to determine if the high-sodium meal causes greater 1) blood pressure dysregulation 2) decreases in blood vessel function and 3) larger changes in blood sodium in Black compared to White individuals. Other potential questions that could be determined include aging differences or an influence of fitness. The investigators will not exclude other races/ethnicities as the project will also determine the response of other minority groups (e.g. Asian or Latine/Hispanic adults) to a high-salt meal.

Participants will report to the laboratory for four visits. At the first visit, consent for study participation will be obtained and participants will be screened for eligibility. Baseline assessments will be completed which may include fitness testing and body composition assessments. If necessary, these assessments may be completed at a second in-person visit. Participants will then report to the laboratory for two experimental visits. At each visit, participants will consume a randomly assigned meal (i.e., a soup containing either low- or high-salt) and undergo assessments prior to and 30- and 60-minutes after consumption. During the study, all participants will consume both meals, however, the order of exposure will be randomly assigned.

ELIGIBILITY:
Inclusion Criteria:

1. Are between the ages of 19-40.
2. Have blood pressure no higher than 140/90 mmHg.
3. Have a BMI below 35 Kg/m2 (otherwise healthy)
4. Free from metabolic disease (diabetes or renal disease), pulmonary disorders (e.g., COPD, severe asthma, or cystic fibrosis), and cardiovascular disease (peripheral vascular, cardiac, or cerebrovascular).
5. Do not have any precluding medical issues that prevent participants from exercising (i.e., cardiovascular issues, or muscle/joint issues including painful arthritis) or giving blood (e.g., blood thinners).
6. Are not currently smoking, using smokeless tobacco, nor smoked within the past 12 months.

Exclusion Criteria:

1. High blood pressure - greater than 140/90 mmHg
2. Obesity (BMI > 30 kg/m2)
3. History of metabolic disease (diabetes or renal disease), pulmonary disorders (e.g., COPD, severe asthma, or cystic fibrosis), and cardiovascular disease (peripheral vascular, cardiac, or cerebrovascular)
4. Medical issues that prevent safe exercise (i.e., cardiovascular issues, or muscle/joint issues including painful arthritis)
5. Medical issues that prevent giving blood (e.g., blood thinners)
6. Currently smoking, using smokeless tobacco, or vaping (within past 12 monrths)
7. Current pregnancy

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in blood pressure reactivity | Before and one hour after soup, both conditions (high- and low- salt)
  The investigators will measure systolic and diastolic pressure using photoplethysmography at the finger. Systolic and diastolic blood pressure will be assessed at rest and during handgrip exercise. Blood pressure reactivity will be expressed as a change in pressure (mmHg) from baseline to a predetermined time during the stressor (e.g., minute one average and minute two average).

SECONDARY OUTCOMES:
Changes in flow-mediated dilation (FMD) | Before, 30 minutes, and one hour after soup, both conditions (high- and low- salt)
  Flow-mediated vasodilation will be assessed using continuous measures of brachial artery diameter and velocity via duplex Doppler ultrasound (Hitachi Arietta 70). The brachial artery will be imaged in the longitudinal plane proximal to the medial epicondyle using a high-frequency (6-12 MHz) linear-array probe. The ultrasound probe will be stabilized using a custom-built clamp. Shear rate (sec-1) will be calculated as [(blood flow velocity (cm*s-1) *4)/blood vessel diameter (mm)] The image will be recorded throughout a 60-s baseline, a 300-s ischemic stimulus (250 mmHg), and 180 seconds post deflation. FMD will be expressed as % dilation (final diameter-baseline diameter/baseline diameter x 100) and also normalized to the shear stimulus. Allometric scaling will be used if appropriate, including if there are baseline differences in artery diameter by race or condition.

OTHER OUTCOMES:
Changes in indices of arterial stiffness | Before 30 minutes, and one hour after soup, both conditions (high- and low- salt)
  The investigators will use the SphygmoCor XCEL system to assess pulse wave analysis (PWA) and pulse wave velocity (PWV). A high-fidelity strain-gauge transducer is used to obtain the pressure waveform at the carotid and radial pulse. Distances from the carotid artery sampling site to the femoral artery (upper leg instrumented with a thigh cuff for oscillometric sphygmomanometry), and from the carotid artery to the suprasternal notch will be recorded. The investigators will also assess forward and reflective wave magnitudes. PWV will be expressed as cm/s and PWA will be expressed as % (calculated as augmentation pressure divided by the pulse pressure).
Changes in blood biomarkers of nitric oxide bioavailability | Before, 30 minutes, and one hour after soup, both conditions (high- and low- salt)
  The investigators will measure nitric oxide metabolites (nitrate and nitrite nanomolar concentration).
Changes in circulating reactive oxygen species | Before, 30 minutes, and one hour after soup, both conditions (high- and low- salt)
  The investigators will use electron paramagnetic resonance to measure reactive oxygen species (spectra units) in whole blood samples treated with a spin probe.
Changes in plasma sodium | Before, 30 minutes, and one hour after soup, both conditions (high- and low- salt)
  The investigators will measure plasma sodium levels.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Auburn University, Auburn, Alabama
  - Indiana University School of Public Health, Bloomington, Indiana

IPD SHARING:
Plan to Share IPD: Yes
Data with all HIPAA identifiers removed may be shared in future collaborative efforts pending appropriate DMDA approvals
Supporting Information: SAP, ICF, Analytic Code
Time Frame: One year after completion of trial, indefinitely
Access Criteria: A formal plan identifying the intended use fo the data and proper completion of a DMDA and MTA (if needed) with Auburn University and the study PI.

REFERENCES:
- [Background] Wenner MM, Paul EP, Robinson AT, Rose WC, Farquhar WB. Acute NaCl Loading Reveals a Higher Blood Pressure for a Given Serum Sodium Level in African American Compared to Caucasian Adults. Front Physiol. 2018 Oct 1;9:1354. doi: 10.3389/fphys.2018.01354. eCollection 2018. PMID 30327611
- [Background] Babcock MC, Robinson AT, Migdal KU, Watso JC, Wenner MM, Stocker SD, Farquhar WB. Reducing Dietary Sodium to 1000 mg per Day Reduces Neurovascular Transduction Without Stimulating Sympathetic Outflow. Hypertension. 2019 Mar;73(3):587-593. doi: 10.1161/HYPERTENSIONAHA.118.12074. PMID 30661474
- [Background] Dickinson KM, Clifton PM, Burrell LM, Barrett PH, Keogh JB. Postprandial effects of a high salt meal on serum sodium, arterial stiffness, markers of nitric oxide production and markers of endothelial function. Atherosclerosis. 2014 Jan;232(1):211-6. doi: 10.1016/j.atherosclerosis.2013.10.032. Epub 2013 Nov 20. PMID 24401240
- [Background] Migdal KU, Robinson AT, Watso JC, Babcock MC, Serrador JM, Farquhar WB. A high-salt meal does not augment blood pressure responses during maximal exercise. Appl Physiol Nutr Metab. 2020 Feb;45(2):123-128. doi: 10.1139/apnm-2019-0217. Epub 2019 Jun 25. PMID 31238011
- [Derived] Culver MN, Linder BA, Lyons DE, Hutchison ZJ, Garrett CL, McNeil JN, Robinson AT. Do not sleep on vitamin D: vitamin D is associated with sleep variability in apparently healthy adults. Am J Physiol Regul Integr Comp Physiol. 2025 Mar 1;328(3):R262-R273. doi: 10.1152/ajpregu.00168.2024. Epub 2025 Jan 28. PMID 39873709